CLINICAL TRIAL: NCT02939222
Title: Impact of Buccal Bone Thickness on Pathological Peri-implant Bone Loss: A 3-year Prospective Cohort Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18002909-2
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-03

CONDITIONS: Periimplantitis; Oral Surgery
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Routine implant placement (Other): No comparison needed
  Interventions: Device: Implant placement

INTERVENTIONS:
Device: Implant placement — Routine implant placement in the ideal three dimensional implant position

SUMMARY:
Implant placement may trigger bone trauma, which might result in 3-dimensional bone changes. While the process of peri-implant disease is not well understood, implant position within the bony structure might play a role. However, there is no data available on this regard.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years old
* Patients requiring oral rehabilitation through supported prosthesis
* Patients with partial edentulism
* No antibiotic in the last 2 months
* No smoking or smoking <10 cigarettes a day

Exclusion Criteria:

* Systemic diseases uncontrolled
* Implants that because prosthetic characteristics can not be registered probing depth or attachment level appropriately
* Smoking> 10 cigarettes a day
* Pregnant Patients
* Implants that can not be followed in CICOM
* Patients who do not return to regular maintenance therapy every 3-6meses
* Patients who are not controlled periodontal disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10-01; Primary Completion 2021-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of peri-implantitis | 3-years
  Control by routine x-ray peri-implant bone loss

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Implantologia Cirugia Oral y Maxiofacial, Badajoz, Spain